CLINICAL TRIAL: NCT05763147
Title: A Prospective, Multi-center, Randomized, Open Label, Controlled Trial of BD Pre-filled Flush Syringes
Brief Title: Study of BD Pre-filled Flush Syringes in China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MDS-21FLUSHCN01
Record Dates: First submitted 2023-02-28; First posted 2023-03-10 (Actual); Results first posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2023-07

CONDITIONS: Effectiveness and Safety of Pre-filled Flush Syringe

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- PosiFlush™ Pre-filled flush syringes (Suzhou Becton Dickinson Medical Devices Co., Ltd.) (Experimental): PosiFlush™ Pre-filled flush syringes (Suzhou Becton Dickinson Medical Devices Co., Ltd.)
  Interventions: Device: Intravenous Access Device Flushing
- PosiFlush™ Pre-filled Flush Syringes (BD, USA) (Active Comparator): PosiFlush™ Pre-filled Flush Syringes (BD, USA)
  Interventions: Device: Intravenous Access Device Flushing

INTERVENTIONS:
Device: Intravenous Access Device Flushing — locking and flushing the end of catheter line at the intervals of different drug treatment.

SUMMARY:
This study is to compare the BD PosiFlush™ Pre-filled Flush Syringes (manufactured by BD, USA) and evaluate the effectiveness and safety of the pre-filled flush syringes (manufactured by Suzhou Becton Dickinson Medical Devices Co., Ltd.) for locking and flushing the end of catheter line in Chinese popluation.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age >or equal to 18, no limitation on gender; 2. Hospitalized patients; 3. Patients who are anticipated to need or have in situ vascular access catheter devices (This may include: Peripheral Intravenous Catheter (PIVC), Central Venous Catheter (such as peripherally inserted central catheter (PICC)); 4. Patients who are expected to require flushing the vascular access catheter with saline at the beginning, during, or end of infusion therapy, or who require to flush and/or lock vascular access catheters at the beginning, during, the end of drug therapy; 5. Patients who can understand the purpose of the trial, agree to participate in this clinical trial and voluntarily sign the informed consent form.

Exclusion Criteria:

* 1. Patient reports pregnancy or lactation (self-report); 2. Subjects who are known to have blockage or recanalization of vascular access prior to this trial.

  3. Subjects who are known to have uncomfortable symptoms such as redness and pain, or common complication associated with indwelling catheter such as phlebitis and infection at the localized insertion site prior to this trial.

  4. Patient participating in another drug or medical device clinical trial at the time of consent or has participated in a drug or medical device clinical trial within three months before enrollment; 5. Any other situation that, in the option of the Investigator would make the patient considered unfit for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 378 (Actual)
Dates: Start 2022-11-03 (Actual); Primary Completion 2023-12-26 (Actual); Study Completion 2023-12-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chao Chao, Principal Investigator — Beijing Hospital
Locations (3):
- China (3):
  - Beijing Friendship Hospital, Beijing
  - Beijing Hospital, Beijing
  - Beijing Jishuitan Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PosiFlush™ Pre-filled Flush Syringes (Suzhou Becton Dickinson Medical Devices Co., Ltd.) | PosiFlush™ Pre-filled Flush Syringes (BD, USA)
Started | 189 | 189
Completed | 188 | 187
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PosiFlush™ Pre-filled Flush Syringes (Suzhou Becton Dickinson Medical Devices Co., Ltd.) | PosiFlush™ Pre-filled Flush Syringes (BD, USA) | Total
Number analyzed (Participants) | 189 | 189 | 378
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.58 (17.11) | 56.15 (16.87) | 55.86 (16.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 74 | 156
  Male | 107 | 115 | 222
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  China | 189 | 189 | 378
Temperature [Mean (Standard Deviation); unit: ℃] | 36.40 (0.27) | 36.42 (0.30) | 36.41 (0.28)
Pulse [Mean (Standard Deviation); unit: beats per minute] | 76.9 (10.5) | 77.6 (10.8) | 77.3 (10.6)
respiratory rate [Mean (Standard Deviation); unit: breathes per minute] | 18.1 (0.7) | 18.1 (0.5) | 18.1 (0.6)
Systolic blood pressure, SBP [Mean (Standard Deviation); unit: millimeters of mercury (mmHG)] | 122.2 (13.3) | 121.3 (13.6) | 121.8 (13.5)
Diastolic blood pressure, DBP [Mean (Standard Deviation); unit: millimeters of mercury (mmHG)] | 75.0 (8.5) | 74.9 (8.9) | 74.9 (8.7)

OUTCOME MEASURES:

1. Primary Outcome: the Overall Performance for Flushing and / or Locking the Catheters.
Description: Evaluation method:
  Overall performance is assessed by a Nurse, who need to answer the following questions:
  1. Can air in the BD Pre-filled Flush Syringes be expelled successfully?
  2. Can BD Pre-filled Flush Syringes be connected to the catheter smoothly?
  3. Can BD Pre-filled Flush Syringes flush and /or lock the catheter successfully?
  4. Can BD Pre-filled Flush Syringes disconnect from the catheters smoothly?
  5. Any leakage observed at any part of the Flush syringe at any time during the usage?
  Overall performance for flushing and/or locking the catheter is only considered as "success" if:
  Question 1 to 4 answered with "YES", and question 5 answered with "NO".
Time Frame: one hour after treatment
Population: Number of nurses who is 'success' per the evaluation method
  For study group, 1 patient withdrew the study and primary endpoint result was not obtained, the other patient met exclusion criteria 4. For control group, 1 patient withdrew the study and primary endpoint result was not obtained, 2 patient met exclusion criteria 4, and the other 1 patient didn't meet inclusion criteria 4. The 6 patients were not included in PPS.
Measure: Number; unit: participants
Arm/Group | PosiFlush™ Pre-filled Flush Syringes (Suzhou Becton Dickinson Medical Devices Co., Ltd.) | PosiFlush™ Pre-filled Flush Syringes (BD, USA)
Number analyzed (Participants) | 187 | 185
participants | 187 | 185

2. Secondary Outcome: Device Ease of Use
Description: Nurse questionnaire:
  1) Is the plunger easy to push forward when flushing or locking? Score on a 5-point scale: '3' means easy
Time Frame: one hour after treatment
Population: number of nurses who gives '> 3 easy'
  For study group, 1 patient withdrew the study and primary endpoint result was not obtained, the other patient met exclusion criteria 4. For control group, 1 patient withdrew the study and primary endpoint result was not obtained, 2 patient met exclusion criteria 4, and the other 1 patient didn't meet inclusion criteria 4. The 6 patients were not included in PPS.
Measure: Number; unit: participants
Arm/Group | PosiFlush™ Pre-filled Flush Syringes (Suzhou Becton Dickinson Medical Devices Co., Ltd.) | PosiFlush™ Pre-filled Flush Syringes (BD, USA)
Number analyzed (Participants) | 187 | 185
participants | 187 | 185

3. Other Pre Specified Outcome: Number of Adverse Events and Serious Adverse Events
Description: Number of adverse events, Incidence of serious adverse events
Time Frame: 1 hour after treatment
Population: For control group, 2 patients didn't use the study devices and were not included in safety set.
Measure: Count of Participants; unit: Participants
Arm/Group | PosiFlush™ Pre-filled Flush Syringes (Suzhou Becton Dickinson Medical Devices Co., Ltd.) | PosiFlush™ Pre-filled Flush Syringes (BD, USA)
Number analyzed (Participants) | 189 | 187
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: The time frame consists of 3 time periods: From screening period (Day-2,-1,0), flush syringe treatment period (Day1) to follow-up period (Day 1, 1 hour after the flush syringe treatment).
Description: The sponsor shall report to the other clinical trial institutions of medical device, EC, and principal investigators participating in clinical trials, report to the drug regulatory departments of the province, autonomous region and municipality directly under the central government where the sponsor is located.
Arm/Group | PosiFlush™ Pre-filled Flush Syringes (Suzhou Becton Dickinson Medical Devices Co., Ltd.) | PosiFlush™ Pre-filled Flush Syringes (BD, USA)
All-Cause Mortality (participants affected / at risk) | 0/189 | 0/187
Serious Adverse Events (participants affected / at risk) | 0/189 | 0/187
Other Adverse Events (participants affected / at risk) | 1/189 | 0/187
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PosiFlush™ Pre-filled Flush Syringes (Suzhou Becton Dickinson Medical Devices Co., Ltd.) (N=189) | PosiFlush™ Pre-filled Flush Syringes (BD, USA) (N=187)
bleeding spot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — scattered subcutaneous bleeding spots

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol (2022-05-26): https://cdn.clinicaltrials.gov/large-docs/47/NCT05763147/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-23): https://cdn.clinicaltrials.gov/large-docs/47/NCT05763147/SAP_001.pdf
  • Informed Consent Form (2022-06-02): https://cdn.clinicaltrials.gov/large-docs/47/NCT05763147/ICF_002.pdf